CLINICAL TRIAL: NCT02242734
Title: Evaluation of the Effect of Hepatic Impairment on the Pharmacokinetics and Metabolism of Hydrocodone and Its Metabolites Following Administration of Hydrocodone Bitartrate Extended-Release (HC-ER) 20mg Capsules
Brief Title: Pharmacokinetics and Metabolism of Hydrocodone Bitartrate Controlled-Release (HC-CR) in Subjects With Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zogenix, Inc. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ZX002-1001
Record Dates: First submitted 2014-08-19; First posted 2014-09-17 (Estimated); Last update posted 2022-11-10 (Actual); Status verified 2014-09

CONDITIONS: Hepatic Impairment
MeSH Terms: interventions — Hydrocodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mild Hepatic Impairment (Experimental): 20 mg HC-ER
  Interventions: Drug: 20 mg HC-ER
- Moderate Hepatic Impairment (Experimental): 20 mg HC-ER
  Interventions: Drug: 20 mg HC-ER
- No Hepatic Impairment (Experimental): 20 mg HC-ER
  Interventions: Drug: 20 mg HC-ER

INTERVENTIONS:
Drug: 20 mg HC-ER — 1-72 hours
  Other Names: Zohydro ER
  Arms: Mild Hepatic Impairment
Drug: 20 mg HC-ER — 1-72 hours
  Other Names: Zohydro ER
  Arms: Moderate Hepatic Impairment
Drug: 20 mg HC-ER — 1-72 hours
  Other Names: Zohydro ER
  Arms: No Hepatic Impairment

SUMMARY:
Determine the influence of hepatic impairment on the pharmacokinetics and metabolism of Hydrocodone Bitartrate Extended-Release (HC-ER) 20 mg capsules

DETAILED DESCRIPTION:
Pharmacokinetics and relative bioavailability of hydrocodone and its metabolites under fasted conditions

ELIGIBILITY:
Inclusion Criteria:

1. All hepatically-impaired subjects must have meet all of the following inclusion criteria to be enrolled into the study:
2. Male or non-pregnant, non-lactating females. Subjects were aged 18-80 years, inclusive.
3. Subjects must have been a clinical diagnosis of chronic hepatic impairment for duration of at least 6 months classified as mild or moderate as per Child-Pugh classification.
4. Hepatic insufficiency was stable with no acute episodes of illness within the previous 2 months due to deterioration of hepatic function due to any etiology.
5. Female subjects of childbearing potential including those who had a tubal ligation surgery but excluded those who did not have a menstrual period for a minimum of 2 years, had a negative pregnancy test at the Screening and Day -1 visits, and consented to use a medically-acceptable method of contraception throughout the entire study period and for 1 week after the study completed. Medically acceptable methods of contraception included were not limited to abstinence, birth control pills or patches, vaginal rings, diaphragm with vaginal spermicide, Intrauterine Device, and progestin implant or injection (used consistently for 3 months prior to study dosing).
6. Subjects voluntarily provided written informed consent.
7. Subjects, in the Investigator's opinion, were able to complete study procedures

   * All healthy control subjects must have met all hepatic subject inclusion criteria as outlined above with the exception of Inclusion Criteria 3 & 4 above which should be substituted with the following to be enrolled into the study:
   * Must have been matched by age (±10 years) and Body Mass Index (BMI) (± 10% of BMI) with some consideration for race and gender to subjects with hepatic impairment.
   * Were medically healthy with no clinically significant abnormalities in their laboratory profile as deemed by the Investigator.

Exclusion Criteria:

1. Women who were pregnant or breastfeeding
2. Any clinically significant condition that would, in the opinion of the Investigator, preclude study participation
3. Uncontrolled blood pressure, i.e., subject has a sitting systolic blood pressure 180 mmHg or 90 mmHg, and/or a sitting diastolic blood pressure 120 mmHg or 50 mmHg at Screening.
4. Body Mass Index (BMI) >40 kg/m2.
5. Known allergy or hypersensitivity to hydrocodone, or other opioids.
6. Had taken any investigational drug within 30 days prior to the Day 1 Visit or currently enrolled in another investigational drug study.
7. Had used a monoamine oxidase inhibitor within 14 days prior to Day 1.
8. Been taking opioids during the 30 days prior to Day 1 or needing to take opioids during the study period
9. Positive for human immunodeficiency virus (HIV). Healthy control subjects must not have been hepatitis C virus (HCV) positive, hepatically-impaired subjects could be HCV positive but should not have been receiving treatment.
10. History of any illicit substance abuse in the past 2 years or any history of opioid abuse. Subjects should not have been current abusers of alcohol and must have had a negative serum alcohol level at Screening and Day -1.
11. Positive quantitative urine drug screen for illicit drugs, or non-prescribed controlled substances at Screening.
12. Had made a plasma donation within 7 days prior to Day 1.
13. Had made any significant donation or loss of blood within 56 days prior to Day 1.
14. Had taken CYP2D6 and/or CYP3A4 inhibitors within 7 days prior to Day 1 and/or CYP2D6 and/or CYP3A4 inducers within 21 days prior to Day 1.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profile of hydrocodone and its metabolites of 20 mg HC-ER | Day 1-3
  PK parameters including Cmax, Tmax, , AUC 0-t, AUC 0-inf, T1/2 and Kel

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Lasseter, MD, Study Director — Zogenix, Inc.